CLINICAL TRIAL: NCT00251758
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Dexlansoprazole MR (60 mg QD and 90 mg QD) Compared to Placebo on Symptom Relief in Subjects With Symptomatic Non-Erosive Gastroesophageal Reflux Disease (GERD)
Brief Title: Safety and Efficacy of Dexlansoprazole Modified Release Formulation to Treat Heartburn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T-GD04-083; U1111-1114-1811 (Registry Identifier: WHO)
Expanded Access: Available
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Results first posted 2009-03-23 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Non-Erosive Gastroesophageal Reflux Disease(GERD),heartburn
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexlansoprazole MR 60 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Dexlansoprazole MR 90 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexlansoprazole MR — Dexlansoprazole MR 60 mg, capsules, orally, once daily for 4 weeks.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 60 mg QD
Drug: Dexlansoprazole MR — Dexlansoprazole MR 90 mg, capsules, orally, once daily for 4 weeks.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 90 mg QD
Drug: Placebo — Dexlansoprazole placebo-matching capsules, orally, once daily for 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of daily treatment with Dexlansoprazole modified release (MR) (60 mg or 90 mg once daily [QD]) compared to placebo QD in relief of daytime and nighttime heartburn over 4 weeks in subjects with gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, multi-center, placebo-controlled, 3-arm study with a 4 week treatment period. This study will compare the efficacy of daily Dexlansoprazole MR (60 mg and 90 mg) with that of placebo when administered orally as a single daily dose in the morning, before breakfast. The study is designed to evaluate symptom relief in subjects with symptomatic non-erosive GERD. Approximately 450 subjects will be enrolled at approximately 120 U.S. and potentially ex U.S. sites. The study consists of two periods; a Screening Period, which will last a minimum of 7 days and a maximum of 21 days, and a treatment period, which will last 4 weeks.

Because the development plan for Dexlansoprazole MR was revised, the results of 2 identical studies, T-GD04-082 (NCT00241745) and T-GD04-083 (this posting, NCT00251758), were combined and analyzed as a single larger study, referred to as study T-GD04-082. A total of 908 subjects were included in the combined analysis; 416 subjects were enrolled into Study T-GD04-082 and 492 subjects were enrolled into Study T-GD04-083.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Non-Erosive Gastroesophageal Reflux Disease identifying their main symptom as heartburn.

  * History of episodes of heartburn for 6 months or longer prior to screening.
  * History of episodes of heartburn for 4 or more days during the 7 days prior to Day -1 as recorded in the electronic diary.

Exclusion Criteria:

* Use of prescription or non-prescription proton pump inhibitors (PPIs), histamine (H2) receptor antagonists, sucralfate, misoprostol or prokinetics throughout the study
* Erosive Esophagitis seen on endoscopy during study screening.
* Co-existing diseases affecting the esophagus.
* Abnormal laboratory values that suggest significant clinical disease.
* Known acquired immunodeficiency syndrome (AIDS)
* Females pregnant or lactating.
* History of Alcohol abuse.
* History of Cancer within 3 years prior to screening.
* Chronic (>12 doses per month) use of nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclo-oxygenase-2 (COX-2) inhibitors
* Use of antacids (except for study supplied Gelusil® )
* Use of drugs with significant anticholinergic effects
* Need for continuous anticoagulant (blood thinner) therapy
* Endoscopic Barrett's esophagus and/or definite dysplastic changes in the esophagus
* History of dilatation of esophageal strictures, other than a Schatzki's ring (a ring of mucosal tissue near the lower esophageal sphincter)
* Current or historical evidence of Zollinger-Ellison syndrome or other hypersecretory condition
* History of gastric, duodenal or esophageal surgery except simple oversew of an ulcer
* Subjects who, in the opinion of the investigator, are unable to comply with the requirements of the study or are unsuitable for any reason.
* Acute upper gastrointestinal (UGI) hemorrhage within 4 weeks of the Screening endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 908 (Actual)
Dates: Start 2005-12; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (99):
- United States (99):
  - Anniston, Alabama
  - Hueytown, Alabama
  - Huntsville, Alabama
  - Tallassee, Alabama
  - Tuscaloosa, Alabama
  - Tucson, Arizona
  - Little Rock, Arkansas
  - North Little Rock, Arkansas
  - Azusa, California
  - Carmichael, California
  - Cypress, California
  - Fresno, California
  - Los Angeles, California
  - Modesto, California
  - Newport Beach, California
  - Oakland, California
  - Orange, California
  - San Diego, California
  - Santa Maria, California
  - Littleton, Colorado
  - Longmont, Colorado
  - Wheat Ridge, Colorado
  - Bristol, Connecticut
  - Newark, Delaware
  - Fort Myers, Florida
  - Miami, Florida
  - Naples, Florida
  - New Smyrna Beach, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Champaign, Illinois
  - Moline, Illinois
  - North Chicago, Illinois
  - Oak Forest, Illinois
  - Springfield, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Newburgh, Indiana
  - Davenport, Iowa
  - Kansas City, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Chevy Chase, Maryland
  - Prince Frederick, Maryland
  - Jackson, Mississippi
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Egg Harbor, New Jersey
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Akron, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Mogadore, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Mt. Pleasant, South Carolina
  - Sioux Falls, South Dakota
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Kingsport, Tennessee
  - Amarillo, Texas
  - Conroe, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Odessa, Texas
  - Pharr, Texas
  - Seguin, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Lakewood, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- See also: For the Dexilant Package Insert refer to this link — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled at 157 sites in the United States (75 in Study T-GD04-082 [NCT00251745] and 82 in Study T-GD04-083 [this posting, NCT00251758]; date of first dose: 07 December 2005; date of last procedure: 23 May 2006).
Pre-assignment Details: Subjects with endoscopically documented normal esophageal mucosa were enrolled in Dexlansoprazole Modified Release (MR) or Placebo once daily (QD) treatment group; subjects were instructed that lifestyle or behavioral modifications designed to treat their symptoms of Gastroesophageal Reflux Disease (GERD) should not be altered throughout the study.
Groups:
- Placebo QD: Placebo capsules, orally, once daily for up to 4 weeks.
- Dexlansoprazole MR 60 mg QD: Dexlansoprazole MR 60 mg, capsules, orally, once daily for up to 4 weeks.
- Dexlansoprazole MR 90 mg QD: Dexlansoprazole MR 90 mg, capsules, orally, once daily for up to 4 weeks.
Period: Overall Study
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Started | 292 | 312 | 304
Completed | 264 | 285 | 277
Not Completed | 28 | 27 | 27
Not completed — Adverse Event | 7 | 9 | 11
Not completed — Lost to Follow-up | 4 | 2 | 5
Not completed — Withdrawal by Subject | 13 | 7 | 3
Not completed — Unmet Inclusion/Exclusion Criteria | 0 | 6 | 5
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Noncompliant | 0 | 2 | 2
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Per Subject Request | 0 | 0 | 1
Not completed — Per Investigator Request | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD | Total
Number analyzed (Participants) | 292 | 312 | 304 | 908
Age Continuous [Mean (Standard Deviation); unit: years] | 49.0 (13.60) | 48.0 (13.55) | 46.7 (13.64) | 47.9 (13.61)
Age, Customized [Number; unit: participants]
  <45 years | 107 | 125 | 135 | 367
  45 - <65 years | 146 | 155 | 139 | 440
  ≥65 years | 39 | 32 | 30 | 101
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 214 | 213 | 643
  Male | 76 | 98 | 91 | 265
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 8 | 14
  Asian | 9 | 12 | 7 | 28
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 0 | 4
  Black or African American | 34 | 46 | 41 | 121
  White | 240 | 246 | 245 | 731
  More than one race | 5 | 1 | 3 | 9
  Unknown or Not Reported | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 58 | 61 | 179
  Not Hispanic or Latino | 232 | 254 | 243 | 729
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days With Neither Daytime Nor Nighttime Heartburn During Treatment as Assessed by Daily Electronic Diary-Median
Description: The percentage was calculated as the days that were heartburn-free out of the total number of days for which either a daytime or nighttime result was marked.
Time Frame: 4 weeks
Population: Analysis was conducted on an intent-to-treat (ITT) population that included all randomized subjects who received at least 1 dose of study drug and completed at least 1 diary entry for heartburn during treatment. All ITT populations excluded subjects with confirmed Barrett's esophagus and/or definite dysplastic changes.
Measure: Median (Inter-Quartile Range); unit: percentage of days
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 290 | 306 | 298
percentage of days | 17.0 [0.0 to 42.9] | 45.7 [11.1 to 75.0] | 52.7 [15.8 to 79.2]
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — The overall 0.0025 level of significance for the multiple comparisons of each dexlansoprazole MR dose to placebo was controlled using Hochberg's method
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 90 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.15505, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.0025 level without adjustment for multiple comparisons

2. Primary Outcome: Percentage of Days With Neither Daytime Nor Nighttime Heartburn During Treatment as Assessed by Daily Electronic Diary-Mean
Description: as for outcome 1
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 290 | 306 | 298
percentage of days | 24.9 (25.7) | 44.8 (33.8) | 49.1 (34.2)

3. Secondary Outcome: Percentage of Days Without Nighttime Heartburn During Treatment as Assessed by Daily Electronic Diary-Median
Description: The percentage was calculated as the nights that were heartburn-free out of the total number of days for which a nighttime result was marked.
Time Frame: 4 weeks
Population: Analysis was conducted on an ITT population (all randomized subjects who received at least 1 dose of study drug and completed at least 1 diary entry for heartburn during treatment), but excluded subjects without any morning diary entries on Day 1 or later.
Measure: Median (Inter-Quartile Range); unit: percentage of days
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 290 | 306 | 298
percentage of days | 51.0 [18.5 to 81.3] | 72.3 [34.6 to 92.9] | 76.6 [37.0 to 92.6]
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.00001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 90 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 60 mg QD vs Dexlansoprazole MR 90 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.38740, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.0025 level without adjustment for multiple comparisons

4. Secondary Outcome: Percentage of Days Without Nighttime Heartburn During Treatment as Assessed by Daily Electronic Diary-Mean
Description: as for outcome 3
Time Frame: 4 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Number analyzed (Participants) | 290 | 306 | 298
percentage of days | 49.6 (34.1) | 62.0 (34.5) | 64.4 (34.6)

ADVERSE EVENTS:
Arm/Group | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Serious Adverse Events (participants affected / at risk) | 0 | 2 | 1
Other Adverse Events (participants affected / at risk) | 37 | 55 | 54
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Cholecystitis and Cholelithiasis (Hepatobiliary disorders) | 0/292 | 0/312 | 1/304
Non-site Specific Injuries Not Elsewhere Classified (NEC) (Injury, poisoning and procedural complications) | 0/292 | 1/312 | 0/304
Poisoning and Toxicity (Injury, poisoning and procedural complications) | 0/292 | 1/312 | 0/304
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo QD | Dexlansoprazole MR 60 mg QD | Dexlansoprazole MR 90 mg QD
Diarrhoea (Excl Infective) (Gastrointestinal disorders) | 13/292 | 15/312 | 8/304
Gastrointestinal and Abdominal Pains (Excl Oral and Throat) (Gastrointestinal disorders) | 12/292 | 23/312 | 15/304
Nausea and Vomiting Symptoms (Gastrointestinal disorders) | 10/292 | 15/312 | 9/304
Upper Respiratory Tract Infections (Infections and infestations) | 4/292 | 11/312 | 24/304
Headaches NEC (Nervous system disorders) | 15/292 | 13/312 | 11/304

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.